CLINICAL TRIAL: NCT03397043
Title: Protein Requirements in Resistance Trained Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Assistant Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RTF
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Healthy

STUDY DESIGN:
Masking Description: Participants blinded to the protein dose consumed in a given metabolic trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy females (Experimental): All participants receive the intervention: Protein intake (dose). This consists of varying levels of dietary protein intakes, in the form of crystalline amino acids, ranging from 0.2-3.0 g/kg/d
  Interventions: Other: Protein intake (dose)

INTERVENTIONS:
Other: Protein intake (dose) — Protein intake, in the form of crystalline amino acids, will range between 0.2-3.0 g/kg/d

SUMMARY:
In this study, the investigators will use the minimally invasive indicator amino acid oxidation (IAAO) technique to determine protein requirements in weight-trained males. It is hypothesized that the present study will show that protein requirements for weight-trained females are i) greater than the current RDA for non-active individual's comparable estimates, and ii) greater than existing nitrogen balance-based estimates for weight-training individuals

DETAILED DESCRIPTION:
Provided that energy needs are met, the adequate ingestion of dietary amino acids is the most critical nutritional factor to support the optimal remodeling and deposition of lean body mass in individuals of all ages. Current recommendations according to the World Health Organization/Food and Agricultural Organization suggest that daily protein requirements in healthy, non-active adults are 0.8 g/kg/day. However, of primary interest in the present study is the impact that exercise has on the nutritional requirement for dietary amino acids in highly active adults - e.g., individuals performing weight training. Protein requirements for individuals who participate in strength-based exercise training have been suggested to range from 1.2-1.7g protein/kg/day (Rodriguez et al., 2009; Tarnopolsky, 1992; Phillips et al., 2007), which equates to a 50-112% increase from the current RDA. The increased requirement in this population may reflect the requirement for protein to repair/rebuild lean tissues by promoting anabolism (Phillips, 2004). Nutritional requirements for dietary amino acids in adults (both active and non-active) have traditionally been determined utilizing the antiquated and often erroneous nitrogen balance technique (Costaneda et al., 1995; Campbell et al., 1984), which is prone to underestimating protein requirements and therefore provides challenges to making accurate nutritional recommendations (Humayun, Elango, Ball, and Pencharz, 2007). This observation that nitrogen balance underestimates protein requirements in non-active individuals could suggest that protein requirements are much greater than the current WHO/FAO recommendation of 0.8 g/kg/day which was evaluated using the nitrogen balance technique (Rand, Pellett and Young, 2003). As a result, there is a need to re-evaluate recommendations utilizing advanced stable isotope methodology in order to characterize how dietary amino acid needs may be modulated by physical activity. Recent studies using the minimally invasive indicator amino acid oxidation (IAAO) technique have suggested that protein requirements in young men are at least 50% higher than WHO/FAO guidelines based on nitrogen balance data (Humayun, Elango, Ball, and Pencharz, 2007). Furthermore, resistance training has been reported to increase (according to nitrogen balance methodology) protein requirements by up to 75% Tarnopolsky et al., 1992). Therefore, in this study, the investigators will use the IAAO technique to determine protein requirements in weight-trained males. It is hypothesized that the present study will show that protein requirements for weight-trained females are i) greater than the current RDA for non-active individual's comparable estimates, and ii) greater than existing nitrogen balance-based estimates for weight-training individuals.

ELIGIBILITY:
Inclusion Criteria:

* healthy female weight-trained individuals that have trained consistently for >1 year
* complete a physical activity readiness questionnaire (PAR-Q+)
* Train each muscle group (i.e. chest, back, legs) at least twice a week
* Meets strength relative to body weight GUIDELINES adapted from Morton et al., 2016; Chilibeck et al., 1997 (sex specific).

Bench Press:

body weight (kg)*0.7

Leg Press:

body weight (kg)*2.3

Exclusion Criteria:

* sedentary for greater than 1 month in the last 6 months prior to the study
* non-weight stable for the past month
* smoker
* Illicit drug use (e.g. growth hormone, testosterone, etc.)
* Individual plans to increase or decrease body mass in the next 3 months
* Habitually ingests greater than or equal to 3g protein kg/bw/day
* Use of supplements such as creatine and beta-alanine in the last 30 days.
* Hormone-based birth control. Hormonal fluctuations associated with the menstrual cycle have been reported to alter protein metabolism during exercise (Hamadeh, Devries, and Tarnopolsky, 2005) For this reason, the following exclusion criteria will be applied to female participants only: use of birth control and discontinued use within last 3 months
* Inability to adhere to any of the protocol guidelines

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Phenylalanine oxidation | Through study completion: an average of 6 metabolic trials (days), each separated by approximately 1 week
  In µmol/kg/h, the product of F13CO2 and VCO2. F13CO2 is determined via breath enrichment analysis of 13CO2 after 1-13C phenylalanine ingestion, and VCO2 is determined via indirect calorimetry

SECONDARY OUTCOMES:
Phenylalanine rate of appearance | Through study completion: an average of 6 metabolic trials (days), each separated by approximately 1 week
  In µmol/kg/h; calculated from urine analysis of1-13C Phe enrichment
Net protein balance | Through study completion: an average of 6 metabolic trials (days), each separated by approximately 1 week
  In µmol/kg/h; calculated as the difference between whole body net protein synthesis and protein breakdown

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Moore, PhD, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: Undecided